CLINICAL TRIAL: NCT01967979
Title: A Single-Center, Open-Label, One-Sequence, 2-Period, Within-Subject Study in 2 Cohorts to Investigate the Effect of Multiple Doses of Itraconazole (Cohort 1) and Fluoxetine (Cohort 2) on the Pharmacokinetics of a Single Dose of RO5285119 in Healthy Subjects
Brief Title: A Study of the Effect of Multiple Doses of Itraconazole and Fluoxetine on the Pharmacokinetics of a Single Dose of RO5285119 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: BP28977; 2013-003232-76 (EudraCT Number)
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — Fluoxetine; Itraconazole

ARMS (2):
- Cohort 1 (Itraconazole DDI) (Experimental)
  Interventions: Drug: RO5285119; Drug: itraconazole
- Cohort 2 (Fluoxetine DDI) (Experimental)
  Interventions: Drug: RO5285119; Drug: fluoxetine

INTERVENTIONS:
Drug: RO5285119 — Single dose, alone and after repeated administration of itraconazole or fluoxetine
Drug: fluoxetine — Multiple doses
  Arms: Cohort 2 (Fluoxetine DDI)
Drug: itraconazole — Multiple doses
  Arms: Cohort 1 (Itraconazole DDI)

SUMMARY:
This single-center, open-label, one-sequence, 2-period, within-subject study in 2 cohorts will evaluate the effects of multiple doses of itraconazole and fluoxetine on the pharmacokinetics of a single dose of RO5285119 in healthy volunteers. In Cohort 1, subjects will receive a single dose of RO5285119 on Day 1 (Period 1) and, after a wash-out period of 14 days, itraconazole on Days 1-8 of Period 2 with coadministration of RO5285119 on Day 4. In Cohort 2, subjects will receive a single dose of RO5285119 on Day 1 (Period 1) and, after a wash-out period of 14 days, fluoxetine on Days 1-12 of Period 2 with coadministration of RO5285119 on Day 6.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 55 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, and a complete physical examination
* Body mass index (BMI) between 18 to 30 kg/m2 inclusive
* Women must be postmenopausal (for at least 12 months of amenorrhea confirmed by FSH, or for at least 24 months if on hormone replacement therapy) or surgically sterile (absence of ovaries and/or uterus)
* For men with a female partner of child-bearing potential: agreement to use a barrier method of contraception during the treatment period and for at least 3 months after the last dose of study drug

Exclusion Criteria:

* Suspicion of regular consumption of drug of abuse, or history of drug or alcohol abuse
* Positive for hepatitis B, hepatitis C , or HIV infection
* Participation in an investigational drug or device study within 90 days prior to first dosing
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study
* Hypersensitivity to itraconazole, to any of the other ingredients, or to any other triazole antifungal, or any other known contraindications to itraconazole as stated in the SmPC
* Hypersensitivity to fluoxetine or to any of the other ingredients, or any other known contraindications to fluoxetine as stated in the SmPC

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effect of multiple doses of itraconazole and fluoxetine on the pharmacokinetics of a single dose of RO5285119 in healthy volunteers: Maximum concentration (Cmax) / Area under the concentration-time curve (AUC) | up to 5 and 7 days post-dose for cohort 1 and cohort 2, respectively

SECONDARY OUTCOMES:
Safety and tolerability of a single dose of RO5285119 administered in combination with itraconazole (cohort 1) and fluoxetine (cohort 2): Incidence of adverse events | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands